CLINICAL TRIAL: NCT06659380
Title: Modulation of Vaginal Microbiota by Lactobacillus Sp As a Probiotic and Immunomodulatory Agent in Postmenopausal Women with Bacterial Vaginosis
Brief Title: Probiotic Efficacy in Postmenopausal Women with Bacterial Vaginosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Yenti Purnamasari, Principal Investigator, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B3/UN4.6.4.5.31-1/ PP36 / 2024
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Bacterial Vaginosis (BV); Menopause
Keywords: NO
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: All patients will receive Metronidazole antibiotic treatment then blind-randomly be divided into two groups: the treatment group, receiving Floragyn® probiotic tablets (Lapi, Indonesia), and the placebo group, receiving Cal 95® (Lapi, Indonesia). As a control, postmenopausal women without bacterial vaginosis will also be included and receive Floragyn® probiotic tablets only. Patients are assessed at T0, T1 and T7 week.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, investigator, and outcomes assessor are blind to treatment status as well as patients and families.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention (Experimental): This group consist of postmenopausal women diagnosed with bacterial vaginosis. All subjects will receive metronidazole oral 400-500 mg twice daily or 0,75% metronidazole gel 5 grams intravaginally once daily for 5 days, then blind-randomly including to the treatment group and will receive Floragyn® probiotic tablets (Lapi, Indonesia) orally once daily for two weeks.
  Interventions: Dietary Supplement: Metronidazole + Floragyn® probiotic tablets (Lapi, Indonesia)
- Placebo (Placebo Comparator): This group consist of postmenopausal women diagnosed with bacterial vaginosis. All subjects will receive metronidazole oral 400-500 mg twice daily or 0,75% metronidazole gel 5 grams intravaginally once daily for 5 days, then blind-randomly including to the placebo group and will receive Cal95® probiotic tablets (Lapi, Indonesia) orally once daily for two weeks.
  Interventions: Dietary Supplement: Metronidazole + Cal95
- Control (Active Comparator): This group consist of postmenopausal women with no bacterial vaginosis. All subjects will receive Floragyn® probiotic tablets (Lapi, Indonesia) orally once daily for two weeks.
  Interventions: Dietary Supplement: Floragyn® probiotic tablets (Lapi, Indonesia)

INTERVENTIONS:
Dietary Supplement: Metronidazole + Floragyn® probiotic tablets (Lapi, Indonesia) — Metronidazole, sold under the brand name Flagyl among others, is an antibiotic and antiprotozoal medication. It is used either alone or with other antibiotics to treat pelvic inflammatory disease, endocarditis, and bacterial vaginosis. It is effective for dracunculiasis, giardiasis, trichomoniasis, and amebiasis.
  One tablet Floragyn contains Lactobacillus rhamnosus and lactobacillus reuteri, bacteria that are normal flora (good bacteria) of the vagina.
  Arms: Intervention
Dietary Supplement: Metronidazole + Cal95 — Metronidazole, sold under the brand name Flagyl among others, is an antibiotic and antiprotozoal medication. It is used either alone or with other antibiotics to treat pelvic inflammatory disease, endocarditis, and bacterial vaginosis. It is effective for dracunculiasis, giardiasis, trichomoniasis, and amebiasis.
  Cal 95 is a supplement containing multivitamins and minerals including: Calcium, Zinc, Boron and Magnesium. This tablet is used to help meet calcium needs and maintain bone health in menopausal women.
  Arms: Placebo
Dietary Supplement: Floragyn® probiotic tablets (Lapi, Indonesia) — Given to the control group to ensure the ability of probiotics to maintain a healthy vaginal ecosystem and not the opposite.
  Arms: Control

SUMMARY:
This study is a double-blind, randomized, controlled trial (RCT) aimed at evaluating the effects of Lactobacillus sp. probiotic administration on the vaginal microbiota changes in postmenopausal women with bacterial vaginosis and how its affect to immunology profile. Postmenopausal women diagnosed with bacterial vaginosis will be recruited as subjects as long as collected period in this study. All patients will receive Metronidazole antibiotic treatment then blind-randomly be divided into two groups: the treatment group, receiving Floragyn® probiotic tablets (Lapi, Indonesia), and the placebo group, receiving Cal 95® (Lapi, Indonesia). As a control, postmenopausal women without bacterial vaginosis will also be included and receive Floragyn® probiotic tablets only.

DETAILED DESCRIPTION:
Postmenopausal women experience hormonal changes, particularly in estrogen and progesterone levels. The reduction or even cessation of estrogen secretion in postmenopausal women leads to an increased dominance of pathogenic bacteria in the vagina, which during the premenopausal period was inhibited by Lactobacillus sp. The presence of Lactobacillus in the vaginal epithelium acts as a barrier against external pathogens and produces metabolic byproducts that are unfavorable for the growth of other bacteria. The availability of glycogen, which is influenced by estrogen levels, supports the presence of Lactobacillus as an energy source. This association explains why women entering menopause are at increased risk of developing bacterial vaginosis. In addition, it is known that female reproductive hormones regulate both innate and adaptive immune responses and modulate endocrine functions that influence Th1 and Th2 cytokines, suppress excessive inflammation, and restore homeostasis.

This study conduct to investigate the effects of probiotic therapy on the vaginal microbiota changes in menopausal women and its impact on immunological profiles. Administering Lactobacillus sp. probiotics is expected to modulate bacterial growth disrupted during perimenopause and help restore homeostasis.

All postmenopausal women, during sample collected period, who meet the inclusion criteria will be enrolled as research subjects. Initially, vaginal swabs and venous blood samples will be collected to assess the bacterial vaginosis condition and hematological profiles. Once bacterial vaginosis is diagnosed, subjects will receive standard antibiotic therapy, metronidazole oral 400-500 mg twice daily or 0,75% metronidazole gel 5 grams intravaginally once daily for 5 days. 48 hours after antibiotic administration, participants will be randomly divided into two groups: the treatment group, receiving Floragyn® probiotics, and the placebo group, receiving Cal95®. Probiotic or placebo treatment will be administered orally once daily for two weeks. A healthy control group will also be included for comparison and will receive Floragyn® for two weeks.

Four weeks after the last probiotic dose, vaginal swabs and venous blood samples will be collected. The analysis will include pH, glucose, protein levels, and microbiome composition from the vaginal swabs, while venous blood samples will be analyzed for interleukin 6 and 10 levels, as well as inflammatory markers such as platelets, leukocytes, and differential leukocyte counts. The collected data will be analyzed to evaluate microbiome alterations and inflammatory markers in the treatment and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal with estradiol levels < 25 mg/ml
2. Diagnosed have bacterial vaginosis by an obstetrician and gynecologist

Exclusion Criteria:

1. Medically unable to perform a pap smear examination
2. Experiencing vaginal bleeding of unknown cause
3. Diagnosed or suspected of having a malignant disease
4. Hypersensitivity to the research treatment to be carried out
5. In the last 3 months have received hormone therapy
6. Suffering from acute infectious diseases of the genital organs
7. Using vaginal therapy in any form
8. Suffering from systemic diseases

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Menopausal women with cessation of menopausal cycles for at least 12 months
Enrollment: 12 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Bacterial Vaginosis Status | At 0, 1, and 7 weeks duration of trial
  A health status of woman reproduction diagnosed by nugent score. Nugent score calculations are carried out by looking at bacterial morphology ie Lactobacillus (parallel - sided, gram positive rods), Mobilincus (curved - Gram negative rods), and Gardnerella / Bacteriodes (tiny, gram-variable cocobacilli and rounded, pleomorphic, gram-negative rods with vacuoles). Score 0-3 is normal flora, score 4-6 is intermediate, score 7-10 is bacterial vaginosis.

SECONDARY OUTCOMES:
Total Leukocyte Count | 0 and 7 weeks duration of trial
  Leukocytes function to detect and fight microorganisms or foreign pathogens that can cause disease, such as viruses, fungi, bacteria, and parasites. Increased levels in the body can be a sign of an ongoing inflammatory process. Leukocyte levels in this study were taken using venous blood samples. its level is expressed in units of 10^3/uL and normal values are 4-10 10^3/uL.
Eosinophil Levels | 0 and 7 weeks duration of trial
  Eosinophils are white blood cells that have a primary function in fighting infections and responding to various types of allergens in the body. Eosinophil levels that exceed the normal range should be watched out for because they can indicate an inflammatory disease. Calculation of eosinophil levels is done using venous blood samples. Eosinophil levels are expressed in % units and normal values are 2-4%.
Monocytes level | 0 and 7 weeks duration of trial
  This type of white blood cell functions to capture and fight attacks by fungi, bacteria, viruses, or parasites that enter the body. The normal level of monocytes is around 2-8% of the total number of white blood cells in the body. The sample used for measurement is venous blood.
Lymphocytes level | 0 and 7 weeks duration of trial
  Lymphocytes are white blood cells that play an important role in protecting the body from various infectious diseases. In addition, the level of lymphocytes in the body can also be a sign of certain medical conditions such as infection and inflammation. The normal level of monocytes is around 20-40% of the total number of white blood cells in the body. The sample used for measurement is venous blood.
Interleukin-6 level | 0 and 7 weeks duration of trial
  Interleukin-6 is a cytokine secreted from body tissues into blood plasma, especially in acute or chronic infection phases, and induces an inflammatory response. The sample used to assess interleukin 6 levels is venous blood with a normal value of interleukin 6 in the blood being <4 pg/ml.
Interleukin-10 level | 0 and 7 weeks duration of trial
  Interleukin-10 is a cytokine abundantly secreted by monocytes, which has pleiotropic effects on the immune system and inflammation by inhibiting the activation and effector functions of T cells, monocytes and macrophages. The sample used to assess interleukin 10 levels is venous blood with a normal value of interleukin 10 in the blood being <18 pg/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Alfa Farma Health Clinic, Obstetrics and Gynecology Doctor's Practice., Kendari, South East Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munoz-Barreno A, Cabezas-Mera F, Tejera E, Machado A. Comparative Effectiveness of Treatments for Bacterial Vaginosis: A Network Meta-Analysis. Antibiotics (Basel). 2021 Aug 13;10(8):978. doi: 10.3390/antibiotics10080978. PMID 34439028
- [Background] Cohen CR, Wierzbicki MR, French AL, Morris S, Newmann S, Reno H, Green L, Miller S, Powell J, Parks T, Hemmerling A. Randomized Trial of Lactin-V to Prevent Recurrence of Bacterial Vaginosis. N Engl J Med. 2020 May 14;382(20):1906-1915. doi: 10.1056/NEJMoa1915254. PMID 32402161
- [Background] France M, Alizadeh M, Brown S, Ma B, Ravel J. Towards a deeper understanding of the vaginal microbiota. Nat Microbiol. 2022 Mar;7(3):367-378. doi: 10.1038/s41564-022-01083-2. Epub 2022 Mar 4. PMID 35246662
- [Background] Laniewski P, Herbst-Kralovetz MM. Connecting microbiome and menopause for healthy ageing. Nat Microbiol. 2022 Mar;7(3):354-358. doi: 10.1038/s41564-022-01071-6. PMID 35246661
- [Background] Peacock K, Carlson K, Ketvertis KM. Menopause. 2023 Dec 21. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507826/ PMID 29939603
- [Background] Peebles K, Velloza J, Balkus JE, McClelland RS, Barnabas RV. High Global Burden and Costs of Bacterial Vaginosis: A Systematic Review and Meta-Analysis. Sex Transm Dis. 2019 May;46(5):304-311. doi: 10.1097/OLQ.0000000000000972. PMID 30624309
- See also: Moulton Vaishall R (2018). Sex Hormones in Acquired Immunity and Autoimmune Disease. Frontiers in Immunology. Doi: 10.3389/fimmu.2018.02279 — https://www.frontiersin.org/journals/immunology/articles/10.3389/fimmu.2018.02279/full
- See also: Gliniewicz Karol et al (2019). Comparison of the Vaginal Microbiomes of Premenopausal and Postmenopausal Women. Frontiers in Microbiology. Front Microbiol. 2019;10:193. Doi: 10.3389/fmicb.2019.00193 — https://www.frontiersin.org/journals/microbiology/articles/10.3389/fmicb.2019.00193/full